CLINICAL TRIAL: NCT01966315
Title: The Comparison of Dexmedetomidine and Midazolam for the Sleep of Mechanical Ventilated Intensive Care Unit Patients
Brief Title: The Comparison of Dexmedetomidine and Midazolam for the Sleep in Intensive Care Unit
Status: Terminated | Type: Observational
Why Stopped: The portable PSG machine can not be available any more.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-1307/212-010
Record Dates: First submitted 2013-10-13; First posted 2013-10-21 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2015-12

CONDITIONS: Poor Quality Sleep; Sleep Deprivation; Sleep Arousal Disorders; Delirium
MeSH Terms: conditions — Sleep Deprivation; Sleep Arousal Disorders; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dexmedetomidine group: Dexmedetomidine group is the patients who sedated with dexmedetomidine in intensive care unit. We will randomly allocate using www.randomizer.org.
  They will sedate at the level of RASS -2. The dose of dexmedetomidine will be 0.2-0.7ug/kg/hr.
- Midazolam group: Midazolam group is the patients who sedated with midazolam in intensive care unit. We will randomly allocate using www.randomizer.org.
  They will sedate at the level of RASS -2. The dose of midazolam will be 0.05-0.1 mg/kg/hr.

SUMMARY:
The investigators are going to compare the sleep quality and quantity between dexmedetomidine group and midazolam group using 24 hour polysomnography in critically ill patients. And the investigators also compare the incidence of delirium between the two groups.

DETAILED DESCRIPTION:
Sleep is very important for cognitive and immune function. However, patients in intensive care unit (ICU) have a very poor sleep.

Almost all ventilated patients in intensive care unit (ICU) take a sedative drug. In Korea, most commonly used sedative drugs are dexmedetomidine and midazolam.

The investigators are going to compare the sleep quality and quantity between dexmedetomidine group and midazolam group using 24 hour polysomnography. And the investigators also compare the incidence of delirium between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* sedation patients with dexmedetomidine or midazolam
* over 18 years old

Exclusion Criteria:

* Neurologic disease (stroke, seizure, dementia, hypoxic brain damage)
* Brain infection
* Alcoholics
* Major Depression Disorder, Schizophrenia, Anxiety disorder
* Hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical patients who take a sedative drugs (dexmedetomidine or midazolam).
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The differences of sleep stage, sleep efficiency, arousal index and delirium between dexmedetomidine group and midazolam group | during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Young-Jae Cho, MPH, Study Chair — Division of Pulmonary and Critical Care Medicine, Department of Internal Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Gyeonggi, Republic of Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea